CLINICAL TRIAL: NCT05802706
Title: The Biomechanical Study of Diseased Human Carotid, Femoral and Abdominal Aortic Tissue
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, CNM II Research, University Hospital of Limerick
Other Study IDs: DVS008
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial plaque tissue is retained following the routine endarterectomy procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
This cross-sectional study aims to ascertain the mechanical properties of human carotid/femoral atherosclerotic plaque and abdominal aortic aneurysm tissue and correlate tissue mechanics with novel blood-based biomarkers of cardiovascular calcification.

DETAILED DESCRIPTION:
The study is a non-randomised, controlled, cross-sectional study of diseased human carotid, femoral and abdominal aortic tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with arterial plaque undergoing treatment where the plaque tissue will be surgically removed as per the usual peripheral endarterectomy procedure.
* Able to provide informed consent.

Exclusion Criteria:

* Patients that are unable to give informed consent.
* Seriously ill/unconscious patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for peripheral endarterectomy of the carotid/femoral artery or abdominal aortic aneurysm surgery to remove artery blockage will be invited to take part in this study with no restrictions on patient type.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Calcification feature classification | 10 years
  Identification of particular calcification features of plaque tissue and their influence on mechanical properties which may help clarify the success of stenting in certain patient cohorts compared to others and elucidate the procedural risk of endovascular treatments in plaque with certain calcification types.
Biomarker Analysis | 10 years
  Identification of novel biomarkers of vascular calcification could potentially be used as a predictive tool to highlight those at greatest risk of adverse peri-operative events, to allow for tailored medical treatment approaches and to stream-line patient care and improve patient outcomes.

SECONDARY OUTCOMES:
Cardiovascular Health Critical Mass | 10 years
  To build a critical mass in cardiovascular health, an area of strategic importance for healthcare in Ireland.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Limerick, Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided